CLINICAL TRIAL: NCT03516266
Title: A Cross-sectional Study of Female Pelvic Floor Muscle Function in Chinese Healthy Female
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Liuzhou Maternity and Child Healthcare Hospital (Other); Qingdao Municipal Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Second Affiliated Hospital of Soochow University (Other); Maternity and Child Health Hospital of Changsha (Unknown); Henan Provincial People's Hospital (Other); Huaian Maternal and Child Health Care Hospital (Other); Hunan Provincial Maternal and Child Health Care Hospital (Other); The Fourth Hospital of Shijiazhuang (Other); Shenzhen Luohu District Maternity And Child Healthcare Hospital (Unknown); Second Affiliated Hospital of Wenzhou Medical University (Other); Hubei Shiyan People's Hospital (Unknown); Changzhi Maternity & Child Health Hospital (Other); Maternal and Child Health Care Hospital of Xinjiang Uygur Autonomous Region (Unknown); The First Hospital of Hebei Medical University (Other); Shen-Zhen City Maternity and Child Healthcare Hospital (Other); Dalian Medical University (Other); Maternity and Child Care Center of QinHuangDao City (Unknown); The People's Hospital of Leshan (Other)
Responsible Party: Sponsor
Other Study IDs: JS-1550
Record Dates: First submitted 2018-04-13; First posted 2018-05-04 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Pelvic Floor
Keywords: Pelvic floor muscle strength; Premenopausal nullipara; Childbirth; Postmenopausal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the status of pelvic floor function of healthy female in China, including premenopausal nullipara, premenopausal women with childbirth and postmenopausal women.

DETAILED DESCRIPTION:
This is a cross-sectional survey. The normal physical examination population is divided into three groups,including premenopausal nullipara, premenopausal women with childbirth and postmenopausal women. The pelvic floor muscle function in three groups are evaluated. The modified Oxford Grading Scale and Levator ani testing is used to quantify PFM strength through vaginal palpation. Pelvic floor muscle strength ,endurance, repetition,vaginal contraction pressure and the knack test are evaluated using a PHENIX USB 8 neuromuscular stimulation therapy system (Company: Vivaltis-Electronic Concept Lignon Innovation, Montpellier, France). In six different regions of China according to geographic region (northwest, southwest, north, east, northeast, and central-south China) , 1 or more hospitals in each area are selected as sub-centers, which needs to complete the evaluation of pelvic floor muscle function of 360 cases in 3 groups totally.

ELIGIBILITY:
Inclusion Criteria:

Group A：Premenopausal women without history of abortion or delivery

1. Having sex life and tolerable to vaginal examination
2. Premenopausal women without history of abortion over 16 weeks
3. Premenopausal women without history of childbirth
4. Planning to live locally for a long time

Group B：Premenopausal women with childbirth

1. Having sex life and tolerable to vaginal examination
2. Premenopausal women with childbirth (including cesarean section or natural birth).
3. Planning to live locally for a long time

Group C:Postmenopausal women (over a year, except surgical menopause)

1. Having sex life and tolerable to vaginal examination
2. Postmenopausal women
3. Planning to live locally for a long time

Exclusion Criteria:

1. Incontinence 4 weeks before enrollment
2. History of fecal incontinence
3. Prolapse beyond the level of the hymen
4. History of radical operation of pelvic cavity(cervical cancer,rectal cancer,bladder cancer, ect）
5. History of pelvic radiotherapy
6. History of pelvic floor surgery
7. History of abortion over 16 weeks' pregnancy or in 1 year after delivery
8. Duration of pregnancy
9. Duration of lactation
10. History of hysterectomy
11. Latex allergy
12. Colpitis

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers are divided into three groups, and each clinical center requires at least 120 persons in each group.
  Group A: Premenopausal women without history of abortion or delivery.
  Group B: Premenopausal women with childbirth (including cesarean section or natural birth).
  Group C:Postmenopausal women (except surgical menopause).
Sampling Method: Probability Sample
Enrollment: 7920 (Estimated)
Dates: Start 2018-05-10 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
maximum vaginal contraction pressure | 1 day
  it is measured by manometry, range(80-150cmH2O). The higher values represent better outcomes.

SECONDARY OUTCOMES:
Pelvic floor muscle strength | 1 day
  The modified Oxford Grading Scale is used to quantify PFM strength through vaginal palpation. range(0-5).The higher values represent better outcomes.
  through vaginal palpation.
Pelvic floor muscle strength（repetition） | 1 day
  Levator ani testing is used to quantify PFM strength. range(0-5). The higher values represent better outcomes.
Pelvic floor muscle contraction endurance | 1 day
  muscle contractions maintained for 0 s are defined as grade 0, 1 s as grade I, 2 s as grade II, 3 s as grade III, 4 s as grade IV, and 5 s or longer as grade V. Normal muscles can maintain the contraction for 5 s. range(0-5s). The higher values represent better outcomes.
pelvic organ prolapse quantification | 1 day
  POP-Q is measured when maximum valsalva. range(0-4). stage 0 represents normal.
the knack test | 1 day
  a voluntary PFM contraction before or during coughing. That the contraction could be performed represents normal.
vaginal rest pressure | 1 day
  measure when no vaginal contraction by manometry. range(25-50 cmH2O). the lower and the higher values represent abnormal outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, MD, Principal Investigator — Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences, Beijing, Beiing, China